CLINICAL TRIAL: NCT01405313
Title: Comparison of Modified Adaptive Servoventilation Therapy With Conventional Adaptive Servoventilation Therapy in Patients With Periodic Breathing
Brief Title: Modified Adaptive Servoventilation (ASV) Compared to Conventional ASV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA231210
Record Dates: First submitted 2011-07-21; First posted 2011-07-29 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2012-09

CONDITIONS: Periodic Breathing; Breathing-Related Sleep Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified ASV (Experimental): Modified ASV Enhanced ASV algorithm which includes auto-adjusting expiratory pressure.
  Interventions: Device: Modified Adaptive Servoventilation Device
- Conventional ASV (Active Comparator): Conventional ASV This is the current (predicate) ASV algorithm.
  Interventions: Device: Conventional Adaptive Servoventilation device

INTERVENTIONS:
Device: Modified Adaptive Servoventilation Device — The modified ASV has a greater adaptive response to meet a target ventilation level that is constantly being assessed.
  Other Names: ResMed Enhanced ASV; ASVAuto
  Arms: Modified ASV
Device: Conventional Adaptive Servoventilation device — Pressure support ventilation adapts to meet a target ventilation level that is constantly being assessed.
  Other Names: ResMed AutoSet CS2; ResMed VPAP Adapt SV; ResMed S9 VPAP Adapt
  Arms: Conventional ASV

SUMMARY:
This study will determine if modified adaptive servoventilation (ASV) is as effective as the conventional ASV in treating periodic breathing. The study will determine if the modified ASV reacts appropriately to reduce apneas and hypopneas and provides suitable levels of positive airway pressure compared to conventional ASV.

DETAILED DESCRIPTION:
Adaptive servoventilation (ASV) is a type of non-invasive ventilation which ameliorates central sleep and/or mixed apnea and periodic breathing. Previous studies in the field have shown that treatment of periodic breathing with ASV improves sleep quality and quality of life. In reducing central apneas, ASV reduces overall arousal index, and increases overall slow wave sleep and rapid eye movement (REM) sleep more than oxygen, continuous positive airway pressure or bi-level treatments. ASV can also more effectively reduce central apnea and overall apnea/hypopnea index (AHI) in patients on long-term opiates, and appears to effectively treat Complex Sleep Apnea Syndrome. It is more effective than other forms of non-invasive ventilation for patients with central and/or mixed apnea or periodic breathing, and is better tolerated.

This is a prospective, randomised, crossover, observational study. Subjects will spend one night on conventional ASV and one night on modified ASV with full in-lab polysomnography (PSG) during therapy on both nights.

Objective and subjective parameters will be recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* 21+ years old
* Chronic ResMed ASV therapy patient
* Current ASV therapy for at least 4 weeks
* Able to understand fully the study information and participation requirements
* Provide signed informed consent

Exclusion Criteria:

* Acute cardiac decompensation
* Acute myocardial infarction within last 3 months
* Resuscitation within last 3 months
* Stroke with swallowing disorders or persistent hemiparesis
* Blood pressure test at end expiratory pressure (EEP) 10cmH2O not passed
* Untreated restless legs syndrome
* Alcohol or drug abuse
* Known cancer
* Pregnancy
* Conditions that could interfere with patients participating in and completing the protocol and/or the investigator deems their enrolment unsuitable

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Oldenburg, MD, Principal Investigator — Heart and Diabetes Centre, Ruhr University Bochum
Locations (1):
- Heart and Diabetes Centre, Ruhr University Bochum, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teschler H, Dohring J, Wang YM, Berthon-Jones M. Adaptive pressure support servo-ventilation: a novel treatment for Cheyne-Stokes respiration in heart failure. Am J Respir Crit Care Med. 2001 Aug 15;164(4):614-9. doi: 10.1164/ajrccm.164.4.9908114. PMID 11520725
- [Background] Pepperell JC, Maskell NA, Jones DR, Langford-Wiley BA, Crosthwaite N, Stradling JR, Davies RJ. A randomized controlled trial of adaptive ventilation for Cheyne-Stokes breathing in heart failure. Am J Respir Crit Care Med. 2003 Nov 1;168(9):1109-14. doi: 10.1164/rccm.200212-1476OC. Epub 2003 Aug 19. PMID 12928310
- [Background] Schadlich S, Konigs I, Kalbitz F, Blankenburg T, Busse HJ, Schutte W. [Cardiac efficiency in patients with Cheyne-Stokes respiration as a result of heart insufficiency during long-term nasal respiratory treatment with adaptive servo ventilation (AutoSet CS)]. Z Kardiol. 2004 Jun;93(6):454-62. doi: 10.1007/s00392-004-0083-3. German. PMID 15252739
- [Background] Oldenburg O, Schmidt A, Lamp B, Bitter T, Muntean BG, Langer C, Horstkotte D. Adaptive servoventilation improves cardiac function in patients with chronic heart failure and Cheyne-Stokes respiration. Eur J Heart Fail. 2008 Jun;10(6):581-6. doi: 10.1016/j.ejheart.2008.04.007. Epub 2008 May 16. PMID 18486550
- [Background] Javaheri S, Malik A, Smith J, Chung E. Adaptive pressure support servoventilation: a novel treatment for sleep apnea associated with use of opioids. J Clin Sleep Med. 2008 Aug 15;4(4):305-10. PMID 18763420
- [Result] Oldenburg O, Spiesshofer J, Fox H, Prib N, Horstkotte D. Performance of conventional and enhanced adaptive servoventilation (ASV) in heart failure patients with central sleep apnea who have adapted to conventional ASV. Sleep Breath. 2015 Sep;19(3):795-800. doi: 10.1007/s11325-014-1083-9. Epub 2014 Nov 21. PMID 25413958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinic population already established on ASV therapy.
Pre-assignment Details: All enrolled participants continued through to group assignment.
Groups:
- First Modified ASV Then Conventional ASV: Patients receive Modified ASV algorithm as therapy for 1 night, then Conventional ASV for 1 night
Period: Overall Study
Arm/Group | First Modified ASV Then Conventional ASV
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 21 patients completed the cross over study design
Groups:
- Modified ASV/Conventional ASV: Therapy used was Modified ASV and then Conventional ASV
Arm/Group | Modified ASV/Conventional ASV
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Region of Enrollment [Number; unit: participants]
  Germany | 21

OUTCOME MEASURES:

1. Primary Outcome: Apnea/Hypopnea Index (AHI)
Description: Physiological sleep signals including pulse oximetry (SpO2), respiratory effort and nasal flow, will be recorded, analysed and reported in the form of an index per hour of sleep. Apnea-Hypopnea Index is calculated counting all apneas (reduction of respiratory flow by >90% for at least 10 seconds) plus all hypopneas (reduction of respiratory flow by >30% for at least 10 seconds with a 4% SpO2 reduction) divided by hours of sleep.
Time Frame: One night
Measure: Mean (Standard Deviation); unit: Events per hour
Groups:
- Modified ASV AHI: 1 night of modified ASV therapy with full polysomnography measurements
- Conventional ASV AHI: 1 night of conventional ASV therapy with full polysomnography measurements
Arm/Group | Modified ASV AHI | Conventional ASV AHI
Number analyzed (Participants) | 21 | 21
Events per hour | 3.9 (4.7) | 6.4 (10.9)
Statistical Analysis 1: Comparison: Modified ASV AHI vs Conventional ASV AHI; Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.022, t-test, 1 sided; Mean Difference (Final Values) = 2.5

2. Secondary Outcome: Oxygen Desaturation Index (ODI)
Description: Oxygen desaturation index based on SpO2 measurement of number of dips (number of times per hour of sleep that SpO2 Drops by at least 3% below the basic value) will be recorded, analysed and reported.
Time Frame: One night
Measure: Mean (Standard Deviation); unit: Events per hour
Groups:
- Modified ASV ODI: 1 night of modified ASV therapy with full polysomnography measurements
- Conventional ASV ODI: 1 night of conventional ASV therapy with full polysomnography measurements
Arm/Group | Modified ASV ODI | Conventional ASV ODI
Number analyzed (Participants) | 21 | 21
Events per hour | 5.2 (5.3) | 8.2 (11.8)
Statistical Analysis 1: Comparison: Modified ASV ODI vs Conventional ASV ODI; Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.016, t-test, 1 sided; Mean Difference (Final Values) = 3.00

ADVERSE EVENTS:
Groups:
- Conventional ASV: Intervention was conventional ASV therapy
- Modified ASV: Intervention was modified ASV therapy
Arm/Group | Conventional ASV | Modified ASV
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional ASV (N=21) | Modified ASV (N=21)
Diagnostic Coronary Angiogram (Cardiac disorders) | 1 (1) | 0 (0) — Coronary angiogram performed as patient (NYHA Class III) reported increased dyspnea. No relation to medical device or clinical trial. Expected event because of patient illness.

LIMITATIONS AND CAVEATS:
None to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No